CLINICAL TRIAL: NCT00060853
Title: Reasoning About Social and Economic Knowledge: Identifying the Role of the Human Prefrontal Cortex Using Functional Neuroimaging
Brief Title: Magnetic Resonance Imaging of the Brain in Social and Emotional Reasoning
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030197; 03-N-0197
Record Dates: First submitted 2003-05-14; First posted 2003-05-14 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-05

CONDITIONS: Healthy
Keywords: Amygdala; Orbitofrontal Cortex; Emotion; Cognition; Theory of Mind; Healthy Volunteer; HV

SUMMARY:
This study will use magnetic resonance imaging (MRI) to identify brain regions involved in social and emotional reasoning. It will identify differences in brain activity during task performance between people who have a nervous system illness and those who do not. MRI is a diagnostic tool that uses a strong magnetic field and radio waves to produce images of structural and chemical changes in the brain.

Healthy normal volunteers between 21 and 55 years of age who are right-handed and are native English speakers may be eligible for this study. Candidates will be screened with a medical history, including psychiatric and neurological information.

Participants will be asked to perform social and emotional reasoning tasks, such as sorting and judging rules and rule violations, while undergoing MRI scanning. Some tasks may simply involve viewing items on a screen. Others may involve solving complex problems and responding by pressing buttons. During the scan, the subject lies on a table in a narrow cylinder (the scanner) containing a magnetic field. The scan will last about 2 hours, with subjects asked to lie still for up to 10 minutes at a time.

DETAILED DESCRIPTION:
The purpose of the protocol is to localize the neural regions and systems mediating the forms of knowledge representations hypothesized by the principal investigator to be stored in the human prefrontal cortex. Utilizing a variety of experimental neuropsychological tasks during functional MRI, we will investigate hypotheses regarding the role of the dorsolateral prefrontal cortex in planning, problem solving, economic exchange and reasoning; and the role of ventromedial prefrontal cortex in social cognition and emotional processing. We will ascertain the relationship between so-called [cold] cognitive processes such as planning and [hot] social processes such as mate choice and specific brain regions within the prefrontal cortex. We will also attempt to determine the relationship between non-frontal neural structures involved in emotional expression, such as the amygdala, and those frontal neural structures involved in executive functions that may modulate emotion. In addition, we will attempt to determine the requirements for frontal-parietal versus frontal-temporal network involvement in spatial landmark tasks. The data that we collect in this protocol will be of value in identifying a set of neural regions and distributed networks mediating the forms of knowledge representation stored in the prefrontal cortex. These questions will be addressed over seven separate studies with healthy, normal adult volunteers. The studies will employ within- and between-subject, event-related fMRI designs. The data collected will consist of behavioral measures of cognitive and emotional performance/judgment and corresponding fMRI images.

ELIGIBILITY:
INCLUSION CRITERIA:

In all the studies, subjects will consist of healthy, native English-speaking, right-handed volunteers, as measured by the Edinburgh Handedness Inventory. Subjects will range in age from 21 to 55 years old and they will be included regardless of race.

In studies 4 and 5, equal numbers of males and females will be recruited owing to previous findings of significant sex differences on such tests. In all other studies subjects will be recruited indiscriminately on the basis of sex.

EXCLUSION CRITERIA:

Non-native English speakers and non-right handers will be excluded as mentioned above, as will non-neurologically normal volunteers. Subjects younger than 21 and older than 55 will be excluded. A pregnancy test will be employed with all women of childbearing age. The results must be negative in order to proceed with the MRI.

Subjects with any of the following: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, e.g. metal shavings; insulin pump; or irremovable body piercing will be excluded from the study due to the possible dangerous effects of the magnet upon metal objects in the body.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Start 2003-05; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Belliveau JW, Rosen BR, Kantor HL, Rzedzian RR, Kennedy DN, McKinstry RC, Vevea JM, Cohen MS, Pykett IL, Brady TJ. Functional cerebral imaging by susceptibility-contrast NMR. Magn Reson Med. 1990 Jun;14(3):538-46. doi: 10.1002/mrm.1910140311. PMID 2355835
- [Background] Bergeron C, Pollanen MS, Weyer L, Lang AE. Cortical degeneration in progressive supranuclear palsy. A comparison with cortical-basal ganglionic degeneration. J Neuropathol Exp Neurol. 1997 Jun;56(6):726-34. PMID 9184663